CLINICAL TRIAL: NCT00003669
Title: Phase II Nonrandomized Study of LY353381-HC1 in Patients With Recurrent or Advanced Endometrial Cancer
Brief Title: Hormone Therapy With Arzoxifene Hydrochloride in Treating Women With Recurrent, Advanced, or Metastatic Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 2141; LILLY-H4Z-MC-JWWI; MSKCC-99001; CDR0000066766
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2008-04

CONDITIONS: Endometrial Cancer
Keywords: stage IV endometrial carcinoma; recurrent endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

INTERVENTIONS:
Drug: arzoxifene hydrochloride

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of endometrial cancer cells. Hormone therapy using arzoxifene hydrochloride may fight the endometrial cancer by blocking the use of estrogen by the tumor cells

PURPOSE: This phase II trial is studying how well arzoxifene hydrochloride works in treating women with recurrent, advanced, or metastatic endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective tumor response rate (complete response and partial response) to arzoxifene hydrochloride in patients with recurrent or advanced endometrial cancer. II. Determine the time to progressive disease, time to treatment failure, response duration, and survival in patients with recurrent or advanced endometrial cancer receiving arzoxifene hydrochloride. III. Assess the safety of this treatment in these patients. IV. Measure changes in serum estradiol, follicle stimulating hormone, luteinizing hormone, and sex hormone binding globulin during this treatment in these patients.

OUTLINE: Patients receive oral arzoxifene hydrochloride daily at a fixed dose. Treatment continues in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: Not specified

National Cancer Institute (NCI) registered this trial with Eli Lilly as sponsor. NCI did not update the record when the trial completed. In June 2012, NCI transferred the trial to Lilly's clinicaltrials.gov account and Lilly updated the record with the trial completion date. This trial is not an applicable trial under Food and Drug Administration Amendments Act of 2007 (FDAAA).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent, advanced, or metastatic endometrial cancer not amenable to curative surgery or radiotherapy Patients should have previously undergone radical surgery (minimum of total abdominal hysterectomy and bisalpingoophorectomy), radical radiotherapy, or not be candidate for such procedures Bidimensionally measurable disease by x-ray, CT scan, MRI, or physical exam No papillary serous or clear cell carcinomas of the endometrium Hormone receptor status: Estrogen receptor positive and/or progesterone receptor positive Unknown receptor status patients allowed provided (1) original tumor was well- or moderately-well differentiated (2) had endometrioid histology

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Menopausal status: Not specified Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL (transfusion-independent) Prothrombin time or activated partial thromboplastin time no greater than 1.25 times upper limit of normal (ULN) Hepatic: Bilirubin no greater than 1.5 times normal ALT or AST no greater than 2.5 times ULN (ALT and AST no greater than 5 times ULN in the presence of liver metastases) Renal: Creatinine no greater than 1.5 ULN Other: No other primary malignancy within the past 5 years except adequately treated nonmelanomatous cancer of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for recurrent or metastatic endometrial cancer At least 1 year since prior adjuvant chemotherapy Endocrine therapy: No prior antiestrogen therapy for any stage of endometrial cancer At least 12 months from time of diagnosis since prior raloxifene Prior progesterone treatment allowed Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy and recovered Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-11; Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Huntington Memorial Hospital, Pasadena, California
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Grant/Riverside Methodist Hospitals, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - U.S. Oncology, Houston, Texas